CLINICAL TRIAL: NCT01254994
Title: A Prospective Open Label Control Study to Evaluate the Efficacy and Safety of Entecavir Treatment of Patients With Acute on Chronic Hepatitis B Liver Failure
Brief Title: The Efficacy and Safety of Entecavir Treatment of Patients With Acute on Chronic Hepatitis B Liver Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Lin Bingliang, Third Affiliated Hospital, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Entecavir
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2007-08

CONDITIONS: Liver Failure
Keywords: hepatitis B; acute on chronic liver failure (ACHBLF); entecavir; treatment; predicting
MeSH Terms: conditions — Liver Failure; Hepatitis B; Acute-On-Chronic Liver Failure | interventions — entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Active Comparator): The patients were prescribed the tradition comprehensive medical treatment without entecavir.
  Interventions: Drug: Traditional comprehensive medical treatment
- ETV group (Experimental): All the patients were prescribed the tradition comprehensive medical treatment with entecavir. Entecavir was supplied by the Sino-US Shanghai Squibb Pharmaceutical Co., Ltd. Patients took 0.5 mg entecavir following oral fasting one time per day.
  Interventions: Drug: entecavir

INTERVENTIONS:
Drug: entecavir — Patients in the ETV Group were prescribed 0.5 mg entecavir following oral fasting one time per day.
  Arms: ETV group
Drug: Traditional comprehensive medical treatment — bed rest, sufficient energy and vitamins, reduced glutathione, prostaglandin E1, hepatocyte growth factor (HGF), plasma and albumin, maintenance of water and electrolyte balance, and prevention and treatment of complications, such as infections, hepatic encephalopathy, hemorrhage, hepatorenal syndrome and ascites.
  Arms: Control group

SUMMARY:
To evaluate therapeutic efficacy and predicting factors of entecavir for treating patients with acute on chronic hepatitis B liver failure (ACHBLF). A total of 108 patients with ACHBLF were allocated into either a treatment group (ETV group, n=53) or a control group (n=55). The HBV DNA level, liver function and survival condition of the patients were observed for 48 weeks after enrollment. The factors possibly related to entecavir treatment efficacy were also identified.

ELIGIBILITY:
Inclusion Criteria:

* ACHBLF was diagnosed according to the criteria from the APASL in March 200815 and the program of Prevention and Cure for Viral Hepatitis and Liver Disease amended by the National Symposium on Viral Hepatitis and Liver Disease in September 2000.
* age >18 years
* HBV DNA > 3log10 copy/mL

Exclusion Criteria:

* Pregnant or lactating women.
* Diagnosed or suspected as hepatic carcinoma patients.
* Cases with any serious disease besides CHB, including heart disease, immunologic disease, malignant tumor, etc.
* Patients hypersensitive to nucleoside or nucleoside (acid) analogues or with a history nucleoside antiviral drug treatment.
* A history of drug abuse or alcohol abuse.
* Hepatic encephalopathy degree IV patients who were unable to take orally administered drugs.
* A history of using immunomodulator including steroids
* Conclusive evidence of other co infection s: anti-HAV-IgM positive, anti-HCV positive, anti-HEV positive, anti-HIV positive, autoimmunity liver diseases, Wilson disease, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2007-08; Primary Completion 2009-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
HBV DNA level and liver function | 48 weeks
  HBV DNA level,serum alanine transaminase (ALT), albumin (ALB), total bilirubin (TB), prothrombin time international normalize ratio （INR）， cholesterol (CHOL)

SECONDARY OUTCOMES:
Symptoms,signs and mortality | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lin B Liang, MD, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- See also: The Third Affiliated Hospital of Sun Yat-sen University — http://www.zssy.com.cn